CLINICAL TRIAL: NCT02897869
Title: A Single-center, Open-label, Two Sequence, Crossover Study to Investigate the Interaction Between Amikacin and POL7080 in Healthy Subjects
Brief Title: DDI Study to Investigate Interaction Between Amikacin and POL7080
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: POL7080-009
Record Dates: First submitted 2016-09-02; First posted 2016-09-13 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — murepavadin; Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence 1 (Experimental): Participants will be randomized to one of two treatment sequences. Sequence 1 is: Period 1, POL7080; Period 2, Amikacin; Period 3,POL7080+Amikacin. Each period is separated by a wash-out period of at least 12 days between last dose and start of next treatment.
  Interventions: Drug: POL7080; Drug: Amikacin; Drug: POL7080 + Amikacin
- Treatment sequence 2 (Experimental): Participants will be randomized to one of two treatment sequences. Sequence 1 is: Period 1, Amikacin; Period 2, POL7080; Period 3,POL7080+Amikacin. Each period is separated by a wash-out period of at least 12 days between last dose and start of next treatment.
  Interventions: Drug: POL7080; Drug: Amikacin; Drug: POL7080 + Amikacin

INTERVENTIONS:
Drug: POL7080 — 7 doses of POL7080 alone over 2.5 days
Drug: Amikacin — 3 doses of Amikacin alone over 2.5 days
Drug: POL7080 + Amikacin — 7 doses of POL7080 and 3 doses of Amikacin over 2.5 days

SUMMARY:
Single-center, open-label, 2-sequence, 3-period crossover drug-drug interaction study. Repeated doses of POL7080 and repeated doses of amikacin will be administered alone or combined. In total, 14 subjects will be enrolled to obtain at least 10 evaluable subjects. The study consists of an eligibility screening period, up to 3 treatments periods and a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) subjects between 18 to 55 years of age (inclusive)
* BMI between 18.0-30.0 kg/m2
* Creatinine clearance estimated by Cockroft Gault formula > 80 mL/min and < 160 ml/min (for males), or < 150ml/min (females)
* Non smokers
* Normal audiogram.

Exclusion Criteria:

* History or suspicion of alcohol and/or drug abuse in the last 5 years
* Within 2 months prior to screening: exposure to aminoglycoside antibiotic, chemotherapy, or current use of loop diuretics
* Regular consumption of large amounts of xanthine
* Any medication that inhibits active tubular secretion within 4 weeks prior to first dosing
* Infection with human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV)
* Any signs of renal impairment
* Clinically significant abnormalities (e.g. cardiovascular, laboratory values)
* Clinically significant abnormal ECG

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Multiple dose pharmacokinetics of POL7080 and Amikacin (as appropriate): Peak Plasma Concentration (Cmax) | Up to 4 days for each period
Multiple dose pharmacokinetics of POL7080 and Amikacin (as appropriate):Area under the plasma concentration versus time curve (AUC) | Up to 4 days for each period

SECONDARY OUTCOMES:
Incidence of adverse Events | up to 19 days

CONTACTS AND LOCATIONS:
Locations (1):
- Mönchengladbach, Germany